CLINICAL TRIAL: NCT04654780
Title: Do Taxes on Unhealthy Foods and Subsidies on Healthy Foods Work in Chile ?: Study of Purchasing Decisions and Food Consumption
Brief Title: Study of Purchasing Decisions and Food Consumption: Chile
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Mayor (Other)
Collaborators: Sociedad Chilena de Pediatría (Unknown)
Responsible Party: Principal Investigator, Carolina Vidal, Principal Investigator, Universidad Mayor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FONISSA17I0121
Record Dates: First submitted 2020-11-24; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Evaluate the Effectiveness of Taxes on Unhealthy; Evaluate the Effectiveness Subsidies for Healthy Foods
Keywords: subsidies; taxes; Nutrition policy; Health policy
MeSH Terms: interventions — Taxes

STUDY DESIGN:
Intervention Model Description: Experimental design that simulates real purchase scenarios to evaluate the effects of a fiscal policy on purchase intention. Participants will be randomly assigned to the different intervention and control groups. Each participant must make a purchase in the virtual supermarket.
  The study groups used in this research :
  1. First intervention group (IG1), a "High in" food tax will be applied to study the changes in the purchasing and consumption behavior of the participants in this group. The tax will correspond to a 20% increase over the market price, that is, a tax that reaches the levels recommended by the WHO.
  2. second intervention group (IG2), a subsidy will be applied to fruits and vegetables that means a reduction of 20% in their price, to study the changes in the purchasing and consumption behavior of the participants of said group.
  3. control group (CG) the market or current prices of "High in" foods and subsidies of fruits and vegetables will be applied.
Who Masked: Participant
Masking Description: The participants were masked to the nature of the price sets to which they were assigned (although they were obviously exposed to the prices in the virtual supermarket). They were informed in the informed consent that the study was to evaluate fiscal policies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tax on purchases (Experimental): exposed to high-price purchases of "high in" foods, including sugary drinks.
  Interventions: Behavioral: Taxes
- subsidies on purchases (Experimental): exposed to purchases with prices that consider subsidies in fruits and vegetables.
  Interventions: Behavioral: Subsidies
- Control (Placebo Comparator): It will not be subjected to any intervention and therefore will buy with current or market prices.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Taxes — a "High in" food tax will be applied to study changes in purchasing and consumption behavior of participants in this group. The tax will correspond to a 20% increase over the market price, that is, a tax that reaches the levels recommended by the WHO.
  Arms: tax on purchases
Behavioral: Subsidies — A subsidy will be applied to fruits and vegetables that means a reduction of 20% in their price, to study the changes in purchasing behavior and of the participants of said group.
  Arms: subsidies on purchases
Behavioral: Control — Average or current food prices will apply. Based on the average of the values reported by three supermarkets
  Arms: Control

SUMMARY:
Objective: To evaluate the effectiveness of taxes on unhealthy foods and subsidies for healthy foods in modifying the purchasing and consumption behavior of people in the Metropolitan Region, Chile.

Research hypothesis:

1. The application of a tax that increases the price of "High in" foods by 20% will reduce the purchase and consumption of these foods by 24%.
2. The application of a subsidy that reduces the price of fruits and vegetables by 20% will increase the purchase and consumption of these foods by 17%.
3. People of lower socioeconomic status are more sensitive to price changes than people of higher socioeconomic status.

Methodological design. The research proposal proposes an experimental design that will select the participants from a panel composed of people over 18 years of age, men and women, and of all socioeconomic levels. The methodological design considers a random assignment of the people eligible for the study into 3 groups:

1. First group of intervention (GI1): people who will make their purchases with taxes on food and beverages "High in";
2. Second intervention group (GI2): people who will make their purchases with subsidies for fruits and vegetables;

4. Control group (CG) that will make the purchases with the market prices or currently applied by the supermarkets or purchase scenarios.

Methodology. Participants will make a monthly simulated purchase through a simulated supermarket system with products similar to those found in real supermarkets, including "High in" products and fruits and vegetables. Different prices will be applied to each group depending on the type of food. With the data of simulated purchases, a variation of the demand and by socioeconomic subgroup will be calculated. The results will be compared with the control group.

Expected results. GI1 participants are expected to modify their purchase intention with the "High in" food tax, decreasing the purchase of these products in their simulated purchases, compared to CG participants who will make their simulated purchases without taxes. Likewise, IG2 participants are expected to modify their purchase intention with the fruit and vegetable subsidy, increasing the purchase of these foods, compared to CG participants. Finally, it is assumed that the reduction in simulated purchases of "High in" foods and the increase in simulated purchases of fruits and vegetables vary according to socioeconomic level.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Person responsible for household purchases.
* Living in a household with one or more boys or girls between 2-14 years of age

Exclusion Criteria:

* That in the home there are no dietary restrictions that prevent the development of this research such as eating disorders, food allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-01-05 (Estimated); Study Completion 2021-01-13 (Estimated)

PRIMARY OUTCOMES:
healthiness of the total shopping | one measurement per participant (requested to purchase food for 15 days)
  percent of total unit food items defined as healthy

CONTACTS AND LOCATIONS:
Overall Officials: Carolina G Vidal, Principal Investigator — Escuela de Salud Pública Universidad Mayor, Chile
Locations (1):
- Carolina Gamboa Vidal, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided
It has not been decided yet. However, the project corresponds to a project awarded from public funds. So Fonis will also safeguard the information.
  The results will be published and any information on the project may be requested in a general email from the School of Public Health of the Universidad Mayor (salud.publica@umayor.cl)

REFERENCES:
- [Background] Waterlander WE, Steenhuis IH, de Boer MR, Schuit AJ, Seidell JC. Introducing taxes, subsidies or both: the effects of various food pricing strategies in a web-based supermarket randomized trial. Prev Med. 2012 May;54(5):323-30. doi: 10.1016/j.ypmed.2012.02.009. Epub 2012 Feb 23. PMID 22387008
- [Background] Waterlander WE, Steenhuis IH, de Boer MR, Schuit AJ, Seidell JC. The effects of a 25% discount on fruits and vegetables: results of a randomized trial in a three-dimensional web-based supermarket. Int J Behav Nutr Phys Act. 2012 Feb 8;9:11. doi: 10.1186/1479-5868-9-11. PMID 22316357